CLINICAL TRIAL: NCT01281072
Title: Study To Evaluate Long Term Treatment Effect Of Diapep277® In Patients Who Have Completed Study 901 And Study 910** (Extension To 901)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: DIABETES UNIT (Ambiguous)
Responsible Party: PROP ITAMAR RAZ, HADASSAH MEDICAL CENTER
Allocation: Not Applicable | Model: Single Group
Other Study IDs: 911-DIAPEP277
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Giving a Vaccination in Three Months
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: vaccine

SUMMARY:
Open label study to evaluate long term treatment effect of diapep277.

ELIGIBILITY:
Inclusion Criteria:

1. patient that completed 901 and 910 study.

Exclusion Criteria:

1. cpeptide<0.2

Ages: 20 Years to 50 Years | Sex: All
Age Groups: Adult

PRIMARY OUTCOMES:
c peptide reserve